CLINICAL TRIAL: NCT02252328
Title: Can Simvastatin Significantly Reduce the Amount of Immunosuppressive Medication Required by Patients With Sight Threatening Uveitis? A Phase 2b, Single Site, Randomized, Placebo Controlled, Double Blinded Trial.
Brief Title: Use of Simvastatin as a Steroid Sparing Agent for Uveitis Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14/0172; 2014-003119-13 (EudraCT Number); 14/0172 (Other Grant/Funding Number: The Moulton Trust)
Record Dates: First submitted 2014-09-08; First posted 2014-09-30 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Uveitis
Keywords: Uveitis; Simvastatin; Visual acuity; Corticosteroids; Immunosuppression
MeSH Terms: conditions — Uveitis | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simvastatine (Experimental): Group of patients receiving simvastatin 80mg once daily in addition to standard care
  Interventions: Drug: Simvastatin
- Placebo (Placebo Comparator): Group of patients receiving placebo once daily in addition to standard care
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 80mg once daily
  Arms: Simvastatine
Drug: Placebo — Placebo tablets once daily
  Arms: Placebo

SUMMARY:
The trial will compare the effect on disease control and immunosuppression treatment of adding simvastatin 80mg once daily, over a follow-up and treatment period of 2 years. Patients will be randomised in a 1:1 fashion to standard treatment with placebo or standard treatment with the addition of simvastatin (80mg daily). They will be followed at 3 months intervals for 2 years with a primary end point of mean reduction in corticosteroid dosage at the 12 month follow-up visit.

DETAILED DESCRIPTION:
This is a non-commercial trial to explore the effect of simvastatin 80mg od on the dose of corticosteroids and immunosuppression in patients with sight-threatening uveitis.

In order to detect a clinical effect the study is designed as a double blinded, parallel group, placebo-controlled, randomised trial. Double blinding will be achieved through the use of a placebo as well as a masked clinical assessor.

Based on the reported effect of simvastatin on brain atrophy among multi[le sclerosis patients after 12 months treatment, patients will receive treatment or placebo and will be treated and followed up for 24 months.

Patients randomised to simvastatin will receive a dose of 80mg od. There will be no dose escalation.

Patients will be reviewed every 3 months and will undergo a complete ophthalmic examination with treatment adjustment accordingly.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be >18 years and under 80 years.
2. Both sexes may participate, but, because of possible teratogenicity of simvastatin women may do so only following counselling about the need for adequate contraception.
3. Women of child bearing potential will have to have a negative pregnancy test prior to enrolment.
4. Patients must have been previously diagnosed with intermediate, posterior or panuveitis (as defined by the standardization of uveitis nomenclature group).14
5. Patients must be taking systemic prednisolone 10mg once daily or more.
6. Patients may be treated with or without a second line agent.
7. Patients must be willing and able to provide informed consent

Exclusion Criteria:

1. No associated underlying systemic disease causing the uveitis.
2. Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed until 6 weeks after treatment discontinuation.
3. Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for trial treatment.
4. Females must not be breastfeeding.
5. Patients concomitantly taking ciclosporin, fibrates, amiodarone, amlodipine, verapamil, cytochrome P450 3A4 inhibitors (e.g. itraconazole, ketoconazole, posaconazole, voriconazole), HIV protease inhibitors (e.g. nelfinavir), erythromycin, clarithromycin, telithromycin, nefazodone, gemfibrozil, danazol, fusidic acid, diltiazem or anti-coagulants.
6. Patients will be advised not to drink grapefruit juice during the study.
7. Family history of hereditary muscle disorders.
8. Active Liver disease
9. Severe renal insufficiency.
10. Persistently elevated serum transaminases.
11. Allergies to excipients of simvastatin and placebo
12. Lactose intolerance
13. Involvement in other clinical trials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
1. Change in dose (mg) of prednisolone after 12 months of treatment | 12 months
  To determine whether the mean reduction in prednisolone dosage achieved at 12 months is greater in the simvastatin group compared to the placebo treated group?

SECONDARY OUTCOMES:
The mean reduction in prednisolone achieved at 24 months. | 24 months
The chnage in the number of 2nd-line immunosuppressive drugs at 24 months | 24 months
The number of disease relapses by 24 months | 24 months
Blood cholesterol and lipid levels at 24 months as compared to baseline | 24 months
Change in visual acuity at 12 and 24 months as compared to baseline | 12 and 24 months
Treg and Th17 levels at 12 and 24 months as compared to baseline | 12 and 24 months
Number of patients with adverse events. | 24 months
The change in dose (mg) of 2nd-line immunosuppressive drugs at 24months | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Oren Tomkins-Netzer, MD, PhD, Principal Investigator — University College, London; Sue Lightman, PhD,FRCOphth, Study Chair — University College, London
Locations (1):
- Moorfields Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chataway J, Schuerer N, Alsanousi A, Chan D, MacManus D, Hunter K, Anderson V, Bangham CR, Clegg S, Nielsen C, Fox NC, Wilkie D, Nicholas JM, Calder VL, Greenwood J, Frost C, Nicholas R. Effect of high-dose simvastatin on brain atrophy and disability in secondary progressive multiple sclerosis (MS-STAT): a randomised, placebo-controlled, phase 2 trial. Lancet. 2014 Jun 28;383(9936):2213-21. doi: 10.1016/S0140-6736(13)62242-4. Epub 2014 Mar 19. PMID 24655729